CLINICAL TRIAL: NCT01023724
Title: A Comparison of Post Phacoemulsification Aqueous Flare in Patients Using Ketorolac 0.45% BID and Bromfenac 0.09% BID
Brief Title: A Comparison of Post Phacoemulsification Aqueous Flare in Patients Using Ketorolac 0.45% 2 Times Daily (BID) and Bromfenac 0.09% 2 Times Daily (BID)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bucci Laser Vision Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Frank A. Bucci, Jr., MD, Bucci Laser Vision
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-11-06 1
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-07

CONDITIONS: Post Operative Anterior Chamber Inflammation (Flare)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bromfenac 0.09% (Active Comparator): bromfenac 0.09% drops to be given pre operatively for one day BID, and then postoperatively for 14 days.
  Interventions: Drug: Bromfenac 0.09%
- Acuvail (Active Comparator): Acuvail to be given preoperatively at BID for one day pre op and then post operatively for 14 days.
  Interventions: Drug: Ketorolac Tromethamine 0.45%

INTERVENTIONS:
Drug: Ketorolac Tromethamine 0.45% — Acuvail to be given 1 drop BID for one day prior to surgery and then 1 drop BID post operatively for 14 days.
  Arms: Acuvail
Drug: Bromfenac 0.09% — Drug given one drop BID for one day pre operatively and then BID for 14 days post operatively
  Arms: bromfenac 0.09%

SUMMARY:
Approximately 50 patients undergoing cataract surgery will be randomized in an even allocation (1:1) into two treatment groups, either ketorolac 0.45% BID or bromfenac 0.09% BID. Patients will be instructed to begin dosing study medication in the operative eye the day before surgery and continue dosing until day 14. KOWA flare measurements will be performed at postoperative day one and postoperative day 14. The amount of anterior chamber inflammation (flare) will be objectively measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Scheduled for cataract surgery by phacoemulsification
* Subject must be willing to comply with all study requirements and be willing to give informed consent

Exclusion Criteria:

* Any subject that has a history of uveitis or active iritis
* Subject can have no previous intraocular surgery with the exception of refractive surgery. but not within 6 months
* No ocular use of prostaglandins within 2 weeks of surgery
* Use of oral, injectable or topical steroids,nonsteroidal anti-inflammatory drugs (NSAIDs) or immunosuppressants within 14 days prior to surgery
* Contraindications to NSAIDs
* Active ocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Xibrom: Xibrom drops to be given pre operatively for one day BID, and then postoperatively for 14 days.
Period: Overall Study
Arm/Group | Xibrom | Acuvail
Started | 25 | 25
Completed | 21 | 22
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xibrom | Acuvail | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 19 | 18 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 72 (9) | 71 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Inflammation (Flare)
Description: Anterior chamber flare measured by assessing the number of inflammatory cells in the anterior chamber.
Time Frame: Day 14 of treatment
Measure: Mean (Standard Deviation); unit: photon count per msec (pc/ms)
Arm/Group | Xibrom | Acuvail
Number analyzed (Participants) | 25 | 25
photon count per msec (pc/ms) | 24.48 (21.94) | 21.93 (19.67)

ADVERSE EVENTS:
Arm/Group | Xibrom | Acuvail
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes